CLINICAL TRIAL: NCT00738348
Title: Effect of Perioperative Sivelstat Administration for Liver Resection
Acronym: KMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kochi University (Other)
Responsible Party: Principal Investigator, Takehiro Okabayashi, University, Kochi University
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Prevention
Other Study IDs: ESAR; Kochi University
Record Dates: First submitted 2008-08-18; First posted 2008-08-20 (Estimated); Last update posted 2012-06-08 (Estimated); Status verified 2012-06

CONDITIONS: Liver Diseases
Keywords: surgery
MeSH Terms: conditions — Liver Diseases | interventions — Glucose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 2 (Active Comparator): 250mL of 5% glucose plus 300mg of sivelstat was infected through the vein at 10mL per an hour
  Interventions: Drug: sivelstat
- 1 (Placebo Comparator): 250mL of 5% glucose was injected though the vein at 10mL per an hour
  Interventions: Drug: glucose

INTERVENTIONS:
Drug: sivelstat — sivelstat sodiumhydrate
  Other Names: sivelstat sodiumhydrate, ONO PHARMACEUTICAL CO
  Arms: 2
Drug: glucose — glucose
  Arms: 1

SUMMARY:
It is reported that sivelstat improved and preserved the postoperative renal function in the orthopedic management. Moreover because sivelstat reduced the migration of neutrophil, it improved acute lung injury. During liver resection, Pringle maneuver, clamping the hepatoduodenal ligament, was performed. Pringle maneuver causes reperfusion injury of the liver. We have a hypothesis that sivelstat prevent the warm shock of reperfusion injury of the liver by Pringle maneuver.

DETAILED DESCRIPTION:
Whether the incidence of postoperative morbidities, such as liver failure, renal failure, or congestive heart failure, was reduced by administration of perioperative sivelstat.

ELIGIBILITY:
Inclusion Criteria:

* liver disease which surgical management was indicated

Exclusion Criteria:

* weight loss greater than 10 per cent during the previous 6 months, signs of distant metastasis, or of respiratory, renal or heart disease

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2007-04; Primary Completion 2008-05 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
The incidence of liver damage due to reperfusion injury by Pringle maneuver was measured by several cytokines, including IL-8, IL-6, and HMGB-1. | during hospitalization

SECONDARY OUTCOMES:
The duration of ICU stay and hospital stay, postoperative complications, and the liver damage at 6 POD, measuring hepato-biliary enzyme | during hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Takehiro Okabayashi, MD, PhD, Study Director — Kochi Medical School
Locations (1):
- Kochi Medical School, Kohasu-Okocho, Nankoku, Japan